CLINICAL TRIAL: NCT05531253
Title: An Observational Study of the Relationship Between Respired Gases, Mixed Venous Oxygen Content and Cardiac Output in Mechanically Ventilated Patients Post Cardiac Surgery
Brief Title: Respired Gases in Patients Post Cardiac Surgery
Acronym: REGAPS
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, DrDonTishanWellalagodage, Principal Investigator, University of Oxford
Other Study IDs: 16070; IRAS 306400 (Other: Health Research Authority NHS UK)
Record Dates: First submitted 2022-08-13; First posted 2022-09-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-05

CONDITIONS: Critically Ill; Cardiac Disease; Mitral Valve Disease
Keywords: pulmonary artery catheter; cardiac output; mixed venous oxygen saturation; oxygen consumption; Fick
MeSH Terms: conditions — Critical Illness; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Main cohort: Patients undergoing cardiac surgery who will have a pulmonary artery catheter in-situ at the time of admission to cardiac intensive care postoperatively.
  Interventions: Other: Data collection using the Optical Gas Analyser

INTERVENTIONS:
Other: Data collection using the Optical Gas Analyser — To allow the OGA to acquire certain physiological data during the study it will be necessary to slightly vary the tension of oxygen and carbon dioxide for short periods. The changes involved will be of a lesser magnitude than those often seen due to natural variation over time in critically ill patients. The FiO2 will be increased by around 20% from baseline for several minutes; this is a far more modest increase than is seen with the practice of pre-oxygenation - a transitory increase in fraction of inspired oxygen ( FiO2) to 100% - performed regularly in ICU patients to make certain routine interventions safer. The end-tidal CO2 level will also briefly (1-2 min) be altered by around 1 kPa by transient adjustment of the ventilator settings.

SUMMARY:
Certain diseases relating to the heart can only be definitively treated with surgery. When untreated, these can lead to heart failure with a lack of supply of oxygen-rich blood to the tissues, leading to damage to other organs.

Adults who undergo heart surgery vary greatly in terms of age and relative health. This has significant implications when predicting outcomes in the aftermath of surgery. For example, a 90-year-old man with a variety of comorbidities such as diabetes and high cholesterol who requires a heart valve replacement may have an unfavourable chance of surviving the postoperative period when compared to an 18-year-old woman with no significant medical history undergoing the same procedure.

Almost invariably, patients are admitted to an Intensive Care Unit (ICU) following heart surgery. This is done to facilitate close monitoring of the patients' vital organ functions and to also provide organ support if needed. For the heart, this can include the administration of drugs to help a heart pump forcibly, cause blood vessels to contract and increase blood pressure. Patients who have undergone heart surgery have been placed on a mechanical ventilator, following a tube placed in their windpipe. This form of ventilation often continues in ICU for a period of time, depending on the patient's condition.

One specific type of ICU level monitoring that occurs in patients who have undergone heart surgery is cardiac output monitoring. This involves a thin tube, called a pulmonary artery catheter, that extends from the skin to the heart, via large blood vessels. Cardiac output monitoring is essential in this patient group to guide organ support and to provide information of how well the heart is functioning.

In this observational study, the investigators wish to study patients who have undergone cardiac surgery, are receiving mechanical ventilation and have pulmonary artery catheters inserted. The investigators will collect cardiopulmonary data in these patients and compare these data with values of exhaled and inhaled gases (oxygen and carbon dioxide) over the same time period. This will enable the investigators to investigate the link between cardiopulmonary data and respired gas values.

A better understanding of this link between cardiopulmonary function and oxygen/carbon dioxide values will then inform future studies aiming to determine the effect of various interventions in similar patient groups.

DETAILED DESCRIPTION:
The cardiovascular system of patients undergoing major cardiac surgery may be unstable during the immediate post-operative period. The core interventions employed as part of routine cardiothoracic ICU management of such patients include the administration of fluids and blood, cardiac pacing, and inotropic support. All of these therapies can be guided by a knowledge of the patient's cardiac output and mixed venous oxygen saturation (SvO2). Pulmonary artery catheters provide an invasive approach that allows the measurement of SvO2 (by blood sampling) and cardiac output (by thermodilution).

For any particular patient, there is always a trade-off between the risks of placing a pulmonary artery catheter and the advantages that it brings when managing patients whose cardiovascular status may be unstable. The primary objective of this study is to explore whether continuous measurement of respired gas exchange, when coupled with small (clinically insignificant), transient variations in inspired oxygen and alveolar carbon dioxide, can be used to calculate mixed venous oxygenation and cardiac output without pulmonary artery catheterisation. If so, then this might provide the basis for a non-invasive approach by which estimates of these parameters can be obtained in patients for whom the benefits of a placing a pulmonary artery catheter do not outweigh the risks.

In order to know the mixed venous oxygenation and cardiac output, this study needs to be conducted in patients who are undergoing pulmonary artery catheterisation as part of their standard clinical care. Patients receiving non-invasive cardiac output monitoring will also be considered. In relation to this, in the UK there are approximately 34,000 major cardiac surgeries which take place each year. Major surgeries in this context include, but are not limited to, coronary artery bypass grafting (CABG), valve replacement or repair and proximal aortic repairs or reconstruction. Following surgery, these patients will invariably be admitted to a Cardiothoracic Intensive Care Unit (CTICU) for the purposes of close cardiorespiratory monitoring and intervention. Many of the patients admitted to CTICU in the postoperative period will require cardiac output monitoring as well as SvO2 measurement. To facilitate this pulmonary artery (PA) catheters are inserted in the perioperative period or non-invasive cardiac output monitoring is utilised postoperatively. Standard operating procedures in our CTICU involve mixed venous sampling for continuous mixed venous oximetry and modern thermodilution via heated catheter for cardiac output measurements. Arterial blood gas samples are taken approximately every hour while the patient is mechanically ventilated.

If it is possible to use measurements of respired gas exchange to estimate cardiac output and SvO2, then they have to be very accurate. The opportunity to obtain measurements with the required precision has arisen from the development of technology that uses laser absorption spectroscopy to measure gas exchange: the Optical Gas Analyser (OGA).

The predicted cardiac output and mixed venous oxygenation are obtained from the measurements of gas exchange by non-linear regression. This process involves a computational model of the lung and circulation that, given particular physiological parameter values and an overall respired gas flow, can calculate the respired gas flows for oxygen, carbon dioxide and nitrogen. The process of non-linear regression is used progressively to adjust the physiological parameter values of the model until the calculated respired gas flows from the model closely match those measured with the OGA. The parameters of the model then provide the cardiac output and SvO2.

In terms of comparators, thermodilution via pulmonary artery catheterisation is generally considered the 'practical' gold standard for measurement of cardiac output in clinical practice. These measurements are available from the pulmonary artery catheter as part of standard clinical care. However, the direct Fick approach is really the true gold standard for the measurement of cardiac output. This requires the mixed venous oxygen content (from the pulmonary artery catheter), the arterial oxygen content (from arterial blood gas measurements) and the oxygen consumption of the patient. The last of these measurements is not available clinically, and this makes the direct Fick method impractical for uses in standard clinical care. Of note, the OGA will supply this measurement, and so a calculation of cardiac output by the direct Fick approach should also be possible in this study.

In summary, A better understanding of the cardiorespiratory changes that occur in post cardiac surgery patients undergoing mechanical ventilation will aid future studies seeking to determine how best to guide various forms of therapy. This will, hopefully, lead to better medical care and improved outcomes in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male and female, aged 18 years or above
* Receiving mechanical ventilation via an endotracheal tube in ICU, directly after cardiac surgery
* Have a pulmonary artery catheter in-situ or receive non-invasive cardiac output monitoring

Exclusion Criteria:

• Patient is receiving palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving mechanical ventilation following cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Oxygen (O2) | Up to 12 hours
  Measured from the OGA
Carbon dioxide (CO2) | Up to 12 hours
  Measured from the OGA

SECONDARY OUTCOMES:
Mixed venous oxygen saturation | Up to 12 hours
  Measured from pulmonary artery catheter
Cardiac output | Up to 12 hours
  Measured from pulmonary artery catheter or non-invasive cardiac output monitor

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Robbins, MBBS DPhil, Study Director — University of Oxford
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bersten A. Oh's intensive care manual. Elsevier; 2014.
- [Background] National Institute for Cardiovascular Outcomes Research, 2020. National Adult Cardiac Surgery Audit (NACSA) 2020 Summary Report (2016/17-2018/19 data). Healthcare Quality Improvement Partnership.
- [Background] Savino JS, Hanson CW 3rd, Gardner TJ. Cardiothoracic intensive care: operation and administration. Semin Thorac Cardiovasc Surg. 2000 Oct;12(4):362-70. doi: 10.1053/stcs.2000.20513. PMID 11154731
- [Background] Rodriguez Ziccardi M, Khalid N. Pulmonary Artery Catheterization. 2023 Aug 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482170/ PMID 29489212
- [Background] Cummings B, Hamilton ML, Ciaffoni L, Pragnell TR, Peverall R, Ritchie GA, Hancock G, Robbins PA. Laser-based absorption spectroscopy as a technique for rapid in-line analysis of respired gas concentrations of O2 and CO2. J Appl Physiol (1985). 2011 Jul;111(1):303-7. doi: 10.1152/japplphysiol.00119.2011. Epub 2011 Apr 21. PMID 21512147
- [Background] Ciaffoni L, O'Neill DP, Couper JH, Ritchie GA, Hancock G, Robbins PA. In-airway molecular flow sensing: A new technology for continuous, noninvasive monitoring of oxygen consumption in critical care. Sci Adv. 2016 Aug 10;2(8):e1600560. doi: 10.1126/sciadv.1600560. eCollection 2016 Aug. PMID 27532048
- [Background] Mountain JE, Santer P, O'Neill DP, Smith NMJ, Ciaffoni L, Couper JH, Ritchie GAD, Hancock G, Whiteley JP, Robbins PA. Potential for noninvasive assessment of lung inhomogeneity using highly precise, highly time-resolved measurements of gas exchange. J Appl Physiol (1985). 2018 Mar 1;124(3):615-631. doi: 10.1152/japplphysiol.00745.2017. Epub 2017 Oct 26. PMID 29074714
- [Background] Magor-Elliott SRM, Fullerton CJ, Richmond G, Ritchie GAD, Robbins PA. A dynamic model of the body gas stores for carbon dioxide, oxygen, and inert gases that incorporates circulatory transport delays to and from the lung. J Appl Physiol (1985). 2021 May 1;130(5):1383-1397. doi: 10.1152/japplphysiol.00764.2020. Epub 2021 Jan 21. PMID 33475459
- [Background] Pugsley J, Lerner AB. Cardiac output monitoring: is there a gold standard and how do the newer technologies compare? Semin Cardiothorac Vasc Anesth. 2010 Dec;14(4):274-82. doi: 10.1177/1089253210386386. Epub 2010 Nov 7. PMID 21059611
- [Background] De Maria AN, Raisinghani A. Comparative overview of cardiac output measurement methods: has impedance cardiography come of age? Congest Heart Fail. 2000 Mar-Apr;6(2):60-73. doi: 10.1111/j.1527-5299.2000.80139.x. PMID 12029189
- [Background] Wilkes AR. Heat and moisture exchangers and breathing system filters: their use in anaesthesia and intensive care. Part 2 - practical use, including problems, and their use with paediatric patients. Anaesthesia. 2011 Jan;66(1):40-51. doi: 10.1111/j.1365-2044.2010.06564.x. Epub 2010 Nov 30. PMID 21118189
- [Background] Davis K Jr, Evans SL, Campbell RS, Johannigman JA, Luchette FA, Porembka DT, Branson RD. Prolonged use of heat and moisture exchangers does not affect device efficiency or frequency rate of nosocomial pneumonia. Crit Care Med. 2000 May;28(5):1412-8. doi: 10.1097/00003246-200005000-00026. PMID 10834688
- [Background] Djedaini K, Billiard M, Mier L, Le Bourdelles G, Brun P, Markowicz P, Estagnasie P, Coste F, Boussougant Y, Dreyfuss D. Changing heat and moisture exchangers every 48 hours rather than 24 hours does not affect their efficacy and the incidence of nosocomial pneumonia. Am J Respir Crit Care Med. 1995 Nov;152(5 Pt 1):1562-9. doi: 10.1164/ajrccm.152.5.7582295.
- [Background] Thomachot L, Vialet R, Viguier JM, Sidier B, Roulier P, Martin C. Efficacy of heat and moisture exchangers after changing every 48 hours rather than 24 hours. Crit Care Med. 1998 Mar;26(3):477-81. doi: 10.1097/00003246-199803000-00018. PMID 9504575
- [Background] Thomachot L, Leone M, Razzouk K, Antonini F, Vialet R, Martin C. Randomized clinical trial of extended use of a hydrophobic condenser humidifier: 1 vs. 7 days. Crit Care Med. 2002 Jan;30(1):232-7. doi: 10.1097/00003246-200201000-00033. PMID 11902268
- [Background] Bujang MA, Baharum N. Sample size guideline for correlation analysis. World Journal of Social Science Research . 2016;3(1):37-46